CLINICAL TRIAL: NCT00335543
Title: Preoperative Chemoradiation in Locally Resectable Adenocarcinoma of Pancreatic Head Without Metastasis
Brief Title: Gemcitabine, Cisplatin, and Radiation Therapy Followed By Surgery or Surgery Alone in Treating Patients With Localized Pancreatic Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Interdisziplinare Arbeitsgruppe Gastrointestinaler Tumore der Deutschen Krebsgesellschaft (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: IAGTDK-70-3046-Ho2; CDR0000472206 (Registry Identifier: PDQ (Physician Data Query)); EU-20609; ISRCTN78805636
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Gemcitabine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet know whether giving chemotherapy together with radiation therapy before surgery is more effective than surgery alone in treating pancreatic cancer.

PURPOSE: This randomized phase II trial is studying how well giving gemcitabine and cisplatin together with radiation therapy before surgery works compared to surgery alone in treating patients with localized pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether neoadjuvant chemoradiotherapy comprising gemcitabine hydrochloride, cisplatin, and radiotherapy is better than immediate surgery, in terms of median survival, in patients with locally resectable adenocarcinoma of the pancreatic head.

Secondary

* Compare 3-year survival rate in patients treated with these regimens.
* Compare R0 resection rate in these patients.
* Compare the rate of medium and high toxicity events in these patients.
* Compare the rate of complete and incomplete remission of the tumor as measured by radiographic imaging studies.
* Compare the rate of different regression gradings in resected tumor specimens.
* Compare the quality of life of these patients.

OUTLINE: This is a prospective, randomized, controlled, open-label, multicenter study. Patients are stratified according to participating center and staging laparoscopy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 1 hour on days 1, 8, 22, and 29. Patients also undergo radiotherapy to the tumor and surrounding lymph nodes 5 days a week for 5 weeks followed by 3 more doses of radiotherapy directly to the tumor. Approximately 6 weeks after finishing chemoradiotherapy, patients with no evidence of disease progression undergo surgery to remove the tumor.
* Arm II: Patients undergo surgery to remove the tumor. After surgery, all patients receive adjuvant chemotherapy comprising gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at the end of chemotherapy and before surgery (arm I), and then at 6 weeks, 6 months, 12 months, and 24 months after surgery.

After completion of study treatment, patients are followed every 3 months for 2 years and then at 3 years.

PROJECTED ACCRUAL: A total of 254 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreatic head

  * No tumors of the body or tail, as defined by a tumor lying between the left border of the superior mesenteric vein and the left border of the aorta and/or the left border of the aorta and the hilum of the spleen
* Locally resectable disease by CT scan

  * Major vessels (e.g., portal vein, confluence of mesenteric and splenic vein, superior mesenteric artery, celiac trunk, splenic artery, hepatic artery, or superior mesenteric vein) maximally enclosed ≤ 180° by the tumor
* No infiltration of extrapancreatic organs except the duodenum
* No carcinoma of the ampulla of Vater
* No metastasis
* No peritoneal carcinoma

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Creatinine clearance > 70 mL/min
* Creatinine < 1.5 mg/dL
* Platelet count > 100,000/mm³
* No liver cirrhosis
* Not pregnant
* No New York Heart Association class III or IV heart disease
* No respiratory insufficiency
* No grade III or IV cardiac arrhythmias
* No pathology on EKG
* No other severe cardiopulmonary disease
* No HIV infection
* No other disease that renders the patient unsuitable for one treatment option
* No other malignancy except nonmelanoma skin cancer, carcinoma in situ of the cervix, or other cancer for which the patient was treated with surgery only and has been in complete remission for ≥ 10 years

PRIOR CONCURRENT THERAPY:

* At least 3 months since prior participation in another clinical trial
* No prior or other concurrent treatment for carcinoma of the pancreas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2003-06; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Median survival

SECONDARY OUTCOMES:
3-year survival rate
R0 resection rate
Rate of medium and high toxicity events
Rate of complete and incomplete remission of the tumor as measured by radiographic imaging studies
Rate of different regression gradings in resected tumor specimens
Quality of life before, during, and after therapy

CONTACTS AND LOCATIONS:
Overall Officials: W. Hohenberger, MD, Study Chair — Universitaet Erlangen
Locations (17):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
- Germany (14):
  - Robert Roessle Comprehensive Cancer Center - Charite Campus Buch, Berlin
  - Knappschaft Krankenhaus, Bochum
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Krankenhaus Dresden - Friedrichstadt, Dresden
  - Universitaet Erlangen, Erlangen
  - Arbeitsgruppe Lebermetastasen und Tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie, Frankfurt
  - Klinik am Eichert, Göppingen
  - Chirurgische Universitaetsklinik, Heidelberg
  - Universitaet Leipzig, Leipzig
  - Staedtisches Klinikum Magdeburg, Magdeburg
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen, Tübingen
- Kantonsspital - St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Golcher H, Brunner T, Grabenbauer G, Merkel S, Papadopoulos T, Hohenberger W, Meyer T. Preoperative chemoradiation in adenocarcinoma of the pancreas. A single centre experience advocating a new treatment strategy. Eur J Surg Oncol. 2008 Jul;34(7):756-64. doi: 10.1016/j.ejso.2007.11.012. Epub 2008 Jan 10. PMID 18191528
- [Derived] Golcher H, Brunner TB, Witzigmann H, Marti L, Bechstein WO, Bruns C, Jungnickel H, Schreiber S, Grabenbauer GG, Meyer T, Merkel S, Fietkau R, Hohenberger W. Neoadjuvant chemoradiation therapy with gemcitabine/cisplatin and surgery versus immediate surgery in resectable pancreatic cancer: results of the first prospective randomized phase II trial. Strahlenther Onkol. 2015 Jan;191(1):7-16. doi: 10.1007/s00066-014-0737-7. Epub 2014 Sep 25. PMID 25252602